CLINICAL TRIAL: NCT03196908
Title: Impact of Energy Drink Brands on Heart Rhythm in Healthy Volunteers: A Randomized Controlled Trial
Brief Title: Impact of Energy Drink Brands on Heart Rhythm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Pacific (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 17-109
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Electrical Alternation of Heart; Blood Pressure
Keywords: ECG; Blood Pressure; Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Energy Drink Brand 1 (Experimental): Two 16-oz bottles of Energy Drink Brand 1
  Interventions: Dietary Supplement: Energy Drink Brand 1
- Energy Drink Brand 2 (Experimental): Two 16-oz bottles of Energy Drink Brand 2
  Interventions: Dietary Supplement: Energy Drink Brand 2
- Placebo (Placebo Comparator): Two 16-oz bottles that each contain 390 ml of carbonated water, 20 ml of reconstituted lime juice, and 70 ml of cherry flavoring
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Energy Drink Brand 1 — Two 16-oz containers of Energy Drink Brand 1 consumed in 60 minutes
  Arms: Energy Drink Brand 1
Dietary Supplement: Energy Drink Brand 2 — Two 16-oz containers of Energy Drink Brand 2 consumed in 60 minutes
  Arms: Energy Drink Brand 2
Other: Placebo — Lime juice, water, and cherry flavoring
  Arms: Placebo

SUMMARY:
To assess the cardiac effects of energy drink brands in healthy volunteers

DETAILED DESCRIPTION:
Energy drinks are widely available and globally consumed. There are many brands of energy drinks on the market, and there are differences in the ingredients included. Previous studies have tried to evaluate the safety of energy drinks and have demonstrated a signal for some electrocardiographic (ECG) and hemodynamic effects. However, product related differences need further exploration. This study is designed to assess the effects of 2 different energy drink products on heart rhythm and blood pressure in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults 18 - 40 years old
* Participants must be willing to refrain from caffeine and alcohol use ≥48 hours prior to sessions on Day 1, 8, and 15

Exclusion Criteria:

* Presence of any known medical condition confirmed through participant interview
* QTc interval greater than 450 milliseconds (ms).
* Blood pressure greater than 140/90 mmHg.
* Current smokers
* Concurrent use of prescription, over-the-counter (OTC) or herbal supplements taken on a daily basis (except oral contraceptives).
* Pregnant or currently breast-feeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Corrected QT (QTc) Interval | 4 hours
  Electrocardiograph (ECG) Parameters

SECONDARY OUTCOMES:
QT | 4 hours
  Electrocardiograph (ECG) Parameters
PR | 4 hours
  Electrocardiograph (ECG)Parameters
QRS | 4 hours
  Electrocardiograph (ECG) Parameters
Heart Rate (HR) | 4 hours
  Electrocardiograph (ECG) Parameters
Central blood pressure | 4 hours
  Hemodynamic Parameters
Peripheral blood pressure | 4 hours
  Hemodynamic Parameters

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Shah, PharmD, Principal Investigator — University of the Pacific
Locations (1):
- University of the Pacific, Stockton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah SA, Szeto AH, Farewell R, Shek A, Fan D, Quach KN, Bhattacharyya M, Elmiari J, Chan W, O'Dell K, Nguyen N, McGaughey TJ, Nasir JM, Kaul S. Impact of High Volume Energy Drink Consumption on Electrocardiographic and Blood Pressure Parameters: A Randomized Trial. J Am Heart Assoc. 2019 Jun 4;8(11):e011318. doi: 10.1161/JAHA.118.011318. Epub 2019 May 29. PMID 31137991